CLINICAL TRIAL: NCT03163277
Title: MARaviroc-based Treatment Switch in HIV-positive Patients With HAND: Consequences of Reducing Antiretroviral-associated Neurotoxicity
Brief Title: Using Less Neurotoxic Drugs in Patients With HAND (MARAND-X)
Acronym: (MARAND-X)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sloww accrual and COVID-19 related problems (impossible to perform LPs)
Sponsor: Giovanni Di Perri (Other)
Responsible Party: Sponsor-Investigator, Giovanni Di Perri, Full Professore of Infectious Diseases, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARAND-X
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Hiv; Neurocognitive Dysfunction
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cognition Disorders | interventions — Emtricitabine; Darunavir; Cobicistat; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Continue current antiretroviral regimen
- Reduced Neurotoxicity Arm (Experimental): Emtricitabine plus darunavir/cobicistat plus maraviroc
  Interventions: Drug: emtricitabine, darunavir/cobicistat, maraviroc

INTERVENTIONS:
Drug: emtricitabine, darunavir/cobicistat, maraviroc — Treatment change
  Arms: Reduced Neurotoxicity Arm

SUMMARY:
Neurocognitive disorders are still highly prevalent in the HAART era; despite a dramatic reduction in dementia cases, 15-50% of patients may develop mild or asymptomatic neurocognitive disorders (HIV-associated neurocognitive disorders, HAND).

Among other hypothesis neurotoxicity of antiretrovirals has been postulated but its impact is unknown.

Our hypothesis is that using drugs with reduced in vitro neurotoxicity may improve cognition in HIV-positive patients withHAND.

76 patients with HAND will be randomized to either continue their treatment or switch to emtricitabine, darunavir/cobicistat, maraviroc. Patients will be re-tested 6 months later.

DETAILED DESCRIPTION:
Scientific Rationale for Study / Scientific Study Objectives:

Neurocognitive disorders are still highly prevalent in the HAART era; despite a dramatic reduction in dementia cases, 15-50% of patients may develop mild or asymptomatic neurocognitive disorders (HIV-associated neurocognitive disorders, HAND). It should be highlighted that patients presenting no abnormalities in everyday living activities (asymptomatic neurocognitive disorders, ANI) are at higher risk of worse results in performance-based tests, adherence-based measures and they show a significant risk of progressing to more severe forms of impairment. Excluding significantly confounding comorbidities, several factors have been associated with this neurocognitive decline including a low nadir CD4+ T-lymphocyte count, a high HIV DNA, a lower compartmental viral control, a lower concentration/penetration effectiveness score, a lower efficacy in macrophage-derived cells and antiretroviral-generated neuronal toxicity. However several data point out that vascular abnormalities, very common in HIV-positive patients, may deeply influence neurocognitive disorders development and severity: of note, intima media thickness, a well recognized proxy of systemic atherosclerosis, was associated with HAND.

In case of HAND diagnosis, the only recommended approach is to optimize treatment according to plasma and cerebrospinal fluid (CSF) resistance tests; no strategy is currently suggested in case of suppressed plasma and CSF HIV RNA or in case of low level CSF HIV RNA (without evidence of genotypic resistance). It has been postulated that antiretrovirals may have neurotoxic effects through different mechanisms and such effects might become evident once the beneficial effect of HIV RNA suppression vanishes. Available data suggest that, in vitro, the drugs associated with the least neurotoxic effect were emtricitabine, tenofovir, darunavir and maraviroc. Furthermore, several pieces of evidence and a small randomized trial suggest that maraviroc, in HAART-treated subjects may have beneficial effects in terms of improved neurocognitive function, reduced CSF inflammatory biomarkers and improved MRI markers of neuronal integrity.

No study has so far investigated the effect of using drugs with a low neurotoxic profile in HAART-treated patients with HAND.

Primary objective of the study is the variation in neurocognitive tests (global deficit score), 6 months after treatment switch while secondary objectives include the improvement in other biomarkers of neuronal and vascular integrity.

Methods:

Study Design: Randomized, controlled, pilot study. HIV-positive patients that fulfill the inclusion criteria and that sign the informed consent will be enrolled. Patients will be randomized 1:1 (block randomization) to either continue their treatment or to switch to once-daily emtricitabine (200 mg) plus darunavir/cobicistat (800/150 mg) plus maraviroc (300 mg). A lumbar puncture will be performed 6 months after treatment switch.

Number of Patients: 76 (38 per arm)

ELIGIBILITY:
Inclusion Criteria:

* Age above >18 years;
* Confirmed HIV-positivity;
* Diagnosed with HAND according to the Frascati Criteria;
* On combination antiretroviral treatment;
* No evidence of major resistance associated mutations on previous plasma or CSF samples;
* Plasma HIV RNA <50 copies/mL;
* CSF HIV RNA <50 copies/mL;
* R5-tropic virus as detected by a genotype or phenotype based test before starting HAART or genotype-based test performed on HIV DNA in the previous 12 months;

Exclusion Criteria:

* the use of drugs having major drug-to-drug interaction with maraviroc (for instance rifampicin);
* the use of efavirenz- or darunavir-containing regimens at baseline;
* confounding comorbidities that may influence or affect the diagnosis of HAND including developmental disability, history of traumatic brain injury or of cerebrovascular accident;
* a previous diagnosis of central nervous system opportunistic, autoimmune, neurodegenerative or neoplastic disease;
* severe untreated depression;
* active alcohol or recreational substance abuse (in the previous 3 months);
* not fluent in Italian or unable to complete the neurocognitive tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
6-month variation in global deficit score in NPZ-8 complete neurocognitive tests according to the study arm; | 6 months
  Global deficit score

SECONDARY OUTCOMES:
rs-fMRI | 6 months
  spectroscopic and perfusion markers at MRI as well as the variations in brain connectivity at resting state functional MRI;
EEG-LORETA | 6 months
  electroencephalographic waves using the LORETA software;
CSF HIV RNA | 6 months
  changes in CSF HIV RNA in the two arms
CSF markers | 6 months
  Variation in CSF markers of inflammation or neuronal damage
Blood Brain Barrier Integrity | 6 months
  Variation in CSAR in the two arms
IMT | 6 months
  Variation in carotid intima media thickness in the two arms
TMAO | 6 months
  Variation in trimethylamine-N-oxide in the two arms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stroffolini G, Lazzaro A, Barco A, Pirriatore V, Vai D, Giaccone C, Nigra M, Atzori C, Trunfio M, Bonora S, Di Perri G G, Calcagno A. Changes in Cerebrospinal Fluid, Liver and Intima-media-thickness Biomarkers in Patients with HIV-associated Neurocognitive Disorders Randomized to a Less Neurotoxic Treatment Regimen. J Neuroimmune Pharmacol. 2023 Dec;18(4):551-562. doi: 10.1007/s11481-023-10086-7. Epub 2023 Oct 31. PMID 37906406